CLINICAL TRIAL: NCT05742750
Title: Camrelizumab Combined With Apatinib and Gemcitabine Plus Cisplatin as First-line Therapy for Patients With Inoperable/Metastatic Biliary Tract Cancer (BTC): An Open-label, Single-arm, Single-center, Phase Ib/II Clinical Study
Brief Title: A Phase Ib/II Clinical Study of Camrelizumab and Apatinib Plus GP in the Treatment of Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dong sheng Zhang, Chief physician，professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-OBU-GD-EC-II-005
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Biliary Tract Cancer; Metastatic Biliary Tract Cancer
Keywords: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — camrelizumab; apatinib; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + apatinib and chemotherapies (gemcitabine and cisplatin) (Experimental): Apatinib is a multi-target TKI, which selectively inhibits VEGFR-2.
  Camrelizumabb is a anti-human PD-1 monoclonal antibody.
  Interventions: Drug: Camrelizumab and Apatinib Plus GP

INTERVENTIONS:
Drug: Camrelizumab and Apatinib Plus GP — Patients received apatinib orally at 250 mg once a day irrespective of the patient weight.
  Camrelizumab 200 mg was administered intravenously over 30 minutes every 3 weeks.
  GP chemotherapy: Gemcitabine/Cisplatin (gemcitabine 1000mg/m2 + cisplatin 25mg/m2) will be administered on D1/D8 in every three weeks cycle and up to 8 cycles.
  All patients continued combination treatment until disease progression, unacceptable toxicity, or discontinuation for any reason.
  Other Names: Apatinib (Apatinib Mesylate Tablets, Jiangsu Hengrui Medicine, China); Camrelizumab (Carelizumab for Injection, Jiangsu Hengrui Medicine, China)

SUMMARY:
The objective of this study is to investigate the safety and tolerability of camrelizumab combined with apatinib and chemotherapies (gemcitabine and cisplatin) in patients with advanced biliary tract cancer (BTC).

DETAILED DESCRIPTION:
The study consists of 2 parts, a dose-escalation part (Phase 1) and an expansion part (Phase 2). Both parts will enroll participants with advanced unresectable biliary tract cancer that had not previously treated with systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to comprehend and willing to sign an informed consent form (ICF).
2. Subject must have a pathologically or cytologically confirmed carcinoma (except neuroendocrine) of the biliary tract (intra-hepatic, extra-hepatic (hilar, distal) or gallbladder) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed cholangiocarcinoma/hepatocellular carcinoma histology are excluded.
3. Subject must be 18-75 years of age at the time of signature of the ICF.
4. Subject must have an ECOG performance status of 0-1. Estimated life expectancy no less than 3 months.
5. Subject may not have received prior systemic treatment (chemotherapy or targeted therapy) for advanced BTC. Prior peri-operative chemotherapy is permitted provided it was completed > 6 months from enrollment.
6. Subject must have a lesion that can be accurately assessed at baseline by CT or magnetic resonance imaging (MRI) and is suitable for repeated assessment in accordance with RECIST v1.1.
7. Subject must have normal organ and marrow function as defined below within 14 days of study entry:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥ 75 × 10^9/L, or hemoglobin ≥ 9 g/dL.
   2. International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits. Patients receiving anticoagulation treatment with an agent such as warfarin will not be candidates for the trial. Patients on anticoagulation with low molecular weight or heparinoids are protocol candidates.
   3. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) unless liver metastasis or BTC in which case ≤ 5 × ULN is permitted at the investigator's discretion. Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3 × ULN.
   4. Creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (measured or calculated by Cockcroft and Gault equation).
   5. Baseline left ventricular ejection fraction (LVEF) ≥ 60% measured by echocardiography or Multiple Gated Acquisition Scan (MUGA)

Exclusion Criteria:

* Patients with any of the following were excluded from the study:

  1. Any investigational agents or study drugs from a previous clinical study within 4 weeks of the first dose of study treatment.
  2. Malignancies other than BTC within 5 years prior to study enrollment, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, or breast ductal carcinoma in situ treated surgically with curative intent).
  3. Prior history of brain metastasis (unless previously treated, asymptomatic and stable for at least 3 months) or organ transplant.
  4. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
  5. Active bleeding during the last 4 weeks prior to screening or in the investigator's judgment, the existence of high bleeding tendency lesions such as active gastrointestinal ulcers or prominent esophageal or gastric varices.
  6. Significant cardiovascular disease, including:

     1. Heart disease classified as New York Heart Association class III or IV.
     2. Ongoing uncontrolled hypertension.
     3. History of congenital long QT syndrome.
     4. Ongoing prolonged QT interval corrected for heart rate using Fridericia's method (QTcF) defined as ≥ 470 msec.
  7. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation).
  8. Subjects with atrial fibrillation, that is well controlled with treatment, can be enrolled. Active heart disease including symptomatic heart failure (NYHA class 3 or 4), unstable angina pectoris, uncontrolled cardiac arrhythmia or interstitial lung disease. Prolonged QTcF interval >480 msec.
  9. Ongoing active, uncontrolled infection (must be afebrile for > 48 hours off antibiotics).
  10. With the exception of alopecia, any unresolved toxicities from prior therapy ≥Common Terminology Criteria for Adverse Events (CTCAE) Grade 2.
  11. Pregnancy or breastfeeding. (Women must not be pregnant or breastfeeding since study drugs may harm the fetus or child. All females of childbearing potential [not surgically sterilized and between menarche and 1 year post menopause] must have a negative screening pregnancy test.)
  12. History of human immunodeficiency virus infection.
  13. History of autoimmune disease.
  14. Ascertained hypersensitivity to gemcitabine, cisplatin, camrelizumab or apatinib, or drugs with similar chemical structures, or its inactive components. If there is suspicion that the subject may have an allergy, the subject should be excluded.
  15. Psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements. Judgment by the investigators that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | up to day 22
  Dose limiting toxicities will determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of combination therapy with camrelizumab + apatinib and gemcitabine plus cisplatin. Assessed using the NCI CTCAE v5.0
Recommended phase 2 dose(RP2D) of apatinib | 12 weeks
  To determine a RP2D of apatinib for each population of biliary tract carcinoma subjects.
Objective Response Rate (ORR) | up to 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
Adverse Events (AE) | up to 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.
Disease Control Rate (DCR) | up to 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | up to 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall Survival (OS) | up to 24 months
  OS is the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Zhang, M.D., Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of SunYat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No